CLINICAL TRIAL: NCT01616732
Title: Effect of Testosterone and Diet on Weight
Brief Title: Testosterone and Weight Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Austin Health (Other Government)
Responsible Party: Principal Investigator, Mathis Grossmann, Associate Professor, Austin Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 04495
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-06

CONDITIONS: Obesity in Men
MeSH Terms: interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- testosterone (Active Comparator): against placebo
  Interventions: Drug: Testosterone
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Testosterone — TU im
  Arms: testosterone
Drug: placebo — placebo im
  Arms: placebo

SUMMARY:
The investigators hypothesise that testosterone therapy will synergize with dietary intervention to achieve weight loss. Obese men will receive diet, and be randomised to either testosterone therapy or placebo. Primary outcomes will be weight and body composition.

ELIGIBILITY:
Inclusion Criteria:

* BMI >30

Exclusion Criteria:

* contraindications to testosterone therapy

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-04; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
weight | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Austin Health, Heidelberg, Victoria, Australia

REFERENCES:
- [Derived] Grossmann M, Fui MNT, Nie T, Hoermann R, Clarke MV, Cheung AS, Zajac JD, Davey RA. Changes in white adipose tissue gene expression in a randomized control trial of dieting obese men with lowered serum testosterone alone or in combination with testosterone treatment. Endocrine. 2021 Aug;73(2):463-471. doi: 10.1007/s12020-021-02722-0. Epub 2021 Apr 17. PMID 33864607
- [Derived] Ng Tang Fui M, Prendergast LA, Dupuis P, Raval M, Strauss BJ, Zajac JD, Grossmann M. Effects of testosterone treatment on body fat and lean mass in obese men on a hypocaloric diet: a randomised controlled trial. BMC Med. 2016 Oct 7;14(1):153. doi: 10.1186/s12916-016-0700-9. PMID 27716209